CLINICAL TRIAL: NCT04587531
Title: Understanding Neural Mechanisms Associated With Cranial Electrotherapy Stimulation in Depression
Brief Title: Neural Mechanisms With CES in Depression
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of financing
Sponsor: Electromedical Products International, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UK-MDDEEG
Record Dates: First submitted 2020-10-07; First posted 2020-10-14 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Depression
Keywords: Depression; EEG; Cranial Electrotherapy Stimulation (CES); Alpha-Stim
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: A 6-week, randomized, double-blind, placebo controlled evaluation of efficacy and tolerability of cranial electrotherapy stimulation (CES) for the treatment of adults with depression. EEG readings will evaluate changes in neural signals following CES treatment.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Treatment device will deliver subsensory treatment while the sham device will deliver no treatment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active CES Therapy (Active Comparator): Group receives active treatment for 6 weeks. The intervention used will be cranial electrotherapy stimulation from and Alpha-Stim AID.
  Interventions: Device: Cranial Electrotherapy Stimulation
- Sham CES Therapy (Sham Comparator): Group receives treatment using sham cranial electrotherapy stimulation devices for 6 weeks. No actual treatment will be received. This group will not receive any treatment interventions. The same outcome measures will be used as the treatment group.
  Interventions: Device: Cranial Electrotherapy Stimulation

INTERVENTIONS:
Device: Cranial Electrotherapy Stimulation — Alpha-Stim® AID microcurrent and cranial electrotherapy stimulator will be used. Daily one hour cranial electrotherapy stimulation (CES) treatment using ear clip electrodes with current set at fixed level of 100 uA (a subsensory current level), 0.5 Hertz will be used for active CES treatment group for 6 weeks. For the sham group the Alpha-Stim® AID ear clips will not emit electricity.
  Other Names: Alpha-Stim

SUMMARY:
This study will examine the effect of cranial electrotherapy stimulation (CES) treatment on adults with depression. Scalp based electroencephalogram (EEG) will be utilized to record the brain activity of participants whilst they perform computer based tasks. The aim is to understand if there would be changes in the neural signals following CES.

DETAILED DESCRIPTION:
Patients meeting the inclusion and exclusion criteria and volunteer to participate will be randomly assigned to "Active CES Therapy" and "Sham CES Therapy" groups. Before start of the treatment (active or sham), their medication details or any other form of treatment they are on will be noted down. These patients will be assessed on self-rated Beck Depression Inventory and clinician rated Hamilton Depression Rating Scale. They will be also assessed on neuropsychological functions of attention, executive functions, memory, information processing and emotional processing evaluation using Emotional Test Battery. In addition, 25 patients from each group will undergo EEG recording whilst they perform computer based tasks. These assessments will take place at 4 time points (Pre-treatment, 1 month after treatment, at 3 months, and at 6 months after treatment).

The study will use scalp based electroencephalogram (EEG) to record the brain activity of participants whilst they perform computer based tasks. The aim is to understand if there would be changes in the neural signals following cranial electrotherapy stimulation. Investigators propose to use EEG to investigate if CES therapy will modulate brain responses in a way that leads to better information processing as a mechanism to improve depression. Furthermore, researchers will also investigate changes in EEG based brain connectivity patterns following CES therapy. Therefore, as a mechanism of action for CES therapy could be changes in the functional brain connectivity for efficient information processing. EEG investigation will be helpful to understand this connectivity based mechanism following CES.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, 18 to 65 years of age.
* Each subject must have a level of understanding sufficient to agree to all required tests and examinations and sign an informed consent document.
* Subjects must fulfil ICD-10 criteria for Depressive Episode or Recurrent Depressive Disorders based on clinical assessment and confirmed by short a structured diagnostic interview, MINI.
* Subjects must have an initial score of at least 14 on the BDI at screen and at baseline of study.
* Current depressive episode of at least 4 weeks duration.

Exclusion Criteria:

* Current or past diagnosis of any other major mental disorders (e.g., schizophrenia, bipolar affective disorders)
* Depression with psychotic symptoms
* Dysthymia
* Depression of organic origin
* Substance misuse/ dependence
* Subjects with one or more seizures without a clear and resolved etiology.
* Female subjects who are pregnant.
* Subjects who, in the investigator's judgment, pose a current serious suicidal or homicidal risk

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-07-05 (Actual); Primary Completion 2023-07-17 (Actual); Study Completion 2023-07-17 (Actual)

PRIMARY OUTCOMES:
Change in Electroencephalogram (EEG) pre-and post-treatment | Pre-treatment; 1 month, 3 months, and 6 months post-treatment
  Scalp based EEG to measure changes in neural signals
Change in Beck Depression Inventory score | Week 1 and Week 6
  Self-report standardized measure of depression with scores ranging from 0-63 with higher scores indicating more severe depression.
Change in Hamilton Depression Rating Scale | Week 1 and Week 6
  Clinician rated standardized measure of depression with scores ranging from 0-50, with higher scores indicating more severe depression.

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Kumar, PhD, Principal Investigator — Oxford Brooke University
Locations (1):
- Oxford Brooke University, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Study results will be available via published article. Individual data will be kept confidential by primary investigator